CLINICAL TRIAL: NCT00391703
Title: Assessment of Quadriceps Muscle Electrostimulation Used as an Additional Procedure for Effort Retraining in Patients Suffering From Cystic Fibrosis Associated With Severe Pulmonary Dysfunction
Brief Title: Assessment of Quadriceps Muscle Electrostimulation Used in Patients Suffering From Cystic Fibrosis
Acronym: STIMUCO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrolment difficulties
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: M. Eric Svahn, Clinical Research Department, Grenoble University Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DCIC05/31
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-11

CONDITIONS: Cystic Fibrosis; Mucoviscidosis
Keywords: Cystic fibrosis; mucoviscidosis; electrostimulation; retraining
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Quadriceps electrostimulation program, performed prior to an endurance retraining program using a cycloergometer
  Interventions: Behavioral: Electrostimulation programme: using a cycloergometer
- 2 (Active Comparator): Usual sport activity, performed prior to an endurance retraining program using a cycloergometer
  Interventions: Behavioral: Usual sport activity

INTERVENTIONS:
Behavioral: Electrostimulation programme: using a cycloergometer — Quadriceps electrostimulation programme performed prior to an endurance retraining program using a cycloergometer, for 6 weeks, 60 to 90 minutes by session, 5 to 6 sessions per week
  Arms: 1
Behavioral: Usual sport activity — Usual sport activity performed prior to an endurance retraining program using a cycloergometer
  Arms: 2

SUMMARY:
This is an add-on, randomized, open label, clinical trial that evaluates the use of quadriceps electrostimulation as an additional retraining procedure in patients suffering from cystic fibrosis.

DETAILED DESCRIPTION:
Cystic fibrosis is an autosomal recessive genetic disease due to a mutation of the CFTR protein gene. The CFTR protein transports chloride ions (Cl-) across cell membranes in the lungs, pancreas, digestive tract, reproductive tract, and skin.

CFTR mutation mainly leads to a dysfunction of the pulmonary system and pancreas exocrine function.

Several studies showed that cystic fibrosis commonly induces a reduction of effort tolerance, peripheral muscular strength and work capacity.

Patients suffering from cystic fibrosis with a high endurance capacity have a lower risk of poor prognosis. Those with a severe dyspnea have a higher benefit with a force training or a combined force and endurance training than with endurance training alone.

We propose to study the effect of a quadriceps electrostimulation program, performed prior to an endurance retraining program using a cycloergometer, in patients with cystic fibrosis associated with severe pulmonary dysfunction, to enhance their muscular performance and increase their adherence to the cycloergometer retraining program.

This is a randomized trial with two groups:

Group A: experimental group, twenty patients. Six weeks with electrostimulation program followed by six weeks under a cycloergometer program.

Group B: control group, twenty patients. Six weeks with their usual physical activity followed by six weeks with a cycloergometer program.

The Randomization is stratified on expiratory volume per second. The size of randomization blocks is random because of the open design.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Patient suffering from cystic fibrosis
* Patient has at least three measures of maximum expiratory volume per second <= 45% of the theory among the 6 last measures performed
* Affiliation to French social security
* Capacity to consent

Exclusion Criteria:

* Pregnant women
* Contraindication to application of magnetic field
* Pacemaker
* History of neurosurgical intervention
* Presence of metallic particles near the stimulation site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The six-minute walking distance | 0, 1, 2 months

SECONDARY OUTCOMES:
Cycloergometer test: maximum power, maximum oxygen consumption, minute ventilation | 1 month
Inspiratory reserve volume (IRV), gasometry, dyspnea score | 0, 1, 2 months
Measurement of voluntary maximum force and non cooperative force of the quadriceps | 0, 1, 2 months
Area of quadriceps cross section measured with a scanner | 1, 2 months
Quadriceps muscle mass | 0, 1, 2 months
Quality of life: CFQ14, BDI-TDI questionnaires | 0, 1, 2 months
Compliance with ergocycle rehabilitation | 1 month
HOMA and QUICKI tests | 0, 1, 2 months
Spirometry | 0, 1, 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Claire Cracowski, Dr, Study Director — Pneumology Department of Grenoble University Hospital
Locations (2):
- France (2):
  - Pneumology Department of Grenoble University Hospital, Grenoble, Isere
  - Pneumology Department of Lyon University Hospital, Lyon, Rhone

REFERENCES:
- [Background] Pin I, Grenet D, Scheid P, Domblides P, Stern M, Hubert D. [Specific aspects and care of lung involvement in adults with cystic fibrosis]. Rev Mal Respir. 2000 Aug;17(3 Pt 2):758-78. French. PMID 11076386
- [Background] de Meer K, Gulmans VA, van Der Laag J. Peripheral muscle weakness and exercise capacity in children with cystic fibrosis. Am J Respir Crit Care Med. 1999 Mar;159(3):748-54. doi: 10.1164/ajrccm.159.3.9802112. PMID 10051246
- [Background] Selvadurai HC, Allen J, Sachinwalla T, Macauley J, Blimkie CJ, Van Asperen PP. Muscle function and resting energy expenditure in female athletes with cystic fibrosis. Am J Respir Crit Care Med. 2003 Dec 15;168(12):1476-80. doi: 10.1164/rccm.200303-363OC. Epub 2003 Sep 18. PMID 14500260
- [Background] Lands LC, Heigenhauser GJ, Jones NL. Respiratory and peripheral muscle function in cystic fibrosis. Am Rev Respir Dis. 1993 Apr;147(4):865-9. doi: 10.1164/ajrccm/147.4.865. PMID 8466121
- [Background] Elkin SL, Williams L, Moore M, Hodson ME, Rutherford OM. Relationship of skeletal muscle mass, muscle strength and bone mineral density in adults with cystic fibrosis. Clin Sci (Lond). 2000 Oct;99(4):309-14. PMID 10995596
- [Background] de Meer K, Jeneson JA, Gulmans VA, van der Laag J, Berger R. Efficiency of oxidative work performance of skeletal muscle in patients with cystic fibrosis. Thorax. 1995 Sep;50(9):980-3. doi: 10.1136/thx.50.9.980. PMID 8539680
- [Background] Moser C, Tirakitsoontorn P, Nussbaum E, Newcomb R, Cooper DM. Muscle size and cardiorespiratory response to exercise in cystic fibrosis. Am J Respir Crit Care Med. 2000 Nov;162(5):1823-7. doi: 10.1164/ajrccm.162.5.2003057. PMID 11069820
- [Derived] Vivodtzev I, Decorte N, Wuyam B, Gonnet N, Durieu I, Levy P, Cracowski JL, Cracowski C. Benefits of neuromuscular electrical stimulation prior to endurance training in patients with cystic fibrosis and severe pulmonary dysfunction. Chest. 2013 Feb 1;143(2):485-493. doi: 10.1378/chest.12-0584. PMID 22911373